CLINICAL TRIAL: NCT01631916
Title: Use of Corticosteroids in Children Hospitalized With Community-acquired Pneumonia
Brief Title: Corticosteroids in Community-acquired Pneumonia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to find patients matching inclusion criteria
Sponsor: Hospital General de Niños Pedro de Elizalde (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HGNPE-66-2012
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Community-acquired Pneumonia
Keywords: community-acquired pneumonia; children; respiratory infections
MeSH Terms: conditions — Community-Acquired Pneumonia; Respiratory Tract Infections | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Corticosteroid (Experimental): Dexamethasone 0.6 mg/kg/day or Methylprednisone 1 mg/kg/day
  Interventions: Drug: corticosteroid
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: corticosteroid — Dexamethasone 0.6 mg/kg/day or Methylprednisone 1 mg/kg/day
  Arms: Corticosteroid

SUMMARY:
The purpose of this study is to determine the efficacy of addition of corticosteroid therapy to antibiotics in children hospitalized with community-acquired pneumonia.

The hypothesis is that the use of corticosteroids decreases the length of stay in children hospitalized with community-acquired pneumonia.

DETAILED DESCRIPTION:
Community-acquired pneumonia (CAP) is a common problem in pediatric practice. The lower respiratory tract infections, particularly pneumonia, are a frequent cause of morbidity in children and is the leading cause of mortality in developing countries.

In the last 20 years, despite several research, only a small decrease in morbidity and mortality has been achieved.

Corticosteroids have an immune-modulation effect, not completely elucidated. Most likely, this effect is due to down regulation of pro-inflammatory cytokines.

We postulate that adding corticosteroids to antibiotic treatment of CAP might change the immune response and thereby reduce morbidity, leading to a decrease in patients hospital length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Children hospitalized for community-acquired pneumonia
* 2-18 years old

Exclusion Criteria:

* Pulmonary chronic disease (including asthma)
* Immunodeficiency
* Diseases wich requires corticosteroids therapy (i.e. rheumatic diseases)
* Wheezing in current disease
* Previous hospitalization (14 days prior to admission)
* Pleural effusion on admission
* Malnutrition

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Length of stay | participants will be followed for the duration of hospital stay, usually 5 days

SECONDARY OUTCOMES:
Length of fever | participants will be followed for the duration of hospital stay, usually 5 days
Length of oxygen use | participants will be followed for the duration of hospital stay, usually 5 days

CONTACTS AND LOCATIONS:
Overall Officials: Romina N Chuminatti, MD, Principal Investigator — Hospital General de Niños Pedro de Elizalde
Locations (1):
- Hospital General de NIños Pedro de Elizalde, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Background] Meijvis SC, Hardeman H, Remmelts HH, Heijligenberg R, Rijkers GT, van Velzen-Blad H, Voorn GP, van de Garde EM, Endeman H, Grutters JC, Bos WJ, Biesma DH. Dexamethasone and length of hospital stay in patients with community-acquired pneumonia: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jun 11;377(9782):2023-30. doi: 10.1016/S0140-6736(11)60607-7. Epub 2011 Jun 1. PMID 21636122
- [Background] Confalonieri M, Urbino R, Potena A, Piattella M, Parigi P, Puccio G, Della Porta R, Giorgio C, Blasi F, Umberger R, Meduri GU. Hydrocortisone infusion for severe community-acquired pneumonia: a preliminary randomized study. Am J Respir Crit Care Med. 2005 Feb 1;171(3):242-8. doi: 10.1164/rccm.200406-808OC. Epub 2004 Nov 19. PMID 15557131
- [Background] Weiss AK, Hall M, Lee GE, Kronman MP, Sheffler-Collins S, Shah SS. Adjunct corticosteroids in children hospitalized with community-acquired pneumonia. Pediatrics. 2011 Feb;127(2):e255-63. doi: 10.1542/peds.2010-0983. Epub 2011 Jan 10. PMID 21220397
- [Background] Snijders D, Daniels JM, de Graaff CS, van der Werf TS, Boersma WG. Efficacy of corticosteroids in community-acquired pneumonia: a randomized double-blinded clinical trial. Am J Respir Crit Care Med. 2010 May 1;181(9):975-82. doi: 10.1164/rccm.200905-0808OC. Epub 2010 Feb 4. PMID 20133929